CLINICAL TRIAL: NCT07230002
Title: Effects of Moderate/Severe Traumatic Brain Injury in the Subacute or Chronic Phase on Locomotor Strategies Involved in Navigation in Complex Virtual Environments
Acronym: NAVIGO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pôle Saint Hélier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-A00679-40
Record Dates: First submitted 2025-09-25; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Locomotion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): Patients as well as healthy participants will be asked to perform several exercises under virtual reality conditions. Questionnaires and scales will also be completed by the participants.
  Interventions: Other: Locomotion in a virtual reality setting

INTERVENTIONS:
Other: Locomotion in a virtual reality setting — Patients and participants will be asked to perform several walking/locomotion tasks in a virtual evironment setting. The setting in question is a concert in a parc. The participants will have to walk towards the stage whilst avoiding bumping into "virtual people". A total of 5 different tasks (walking in a straight line, walking between people etc) will be completed for each participant. Different variables will then be recorded and extracted such as walking speed, interpersonnal distances, eye fixation times.

SUMMARY:
While clinical assessment of locomotor function in this population is carried out using tasks involving walking in a straight line without any obstacles, it does not take into account ecological situations (i.e., situations comparable to real-life situations) in which the person interacts with their environment, such as walking down a street with other pedestrians, which is fundamental to everyday life. This research therefore aims to study the social navigation skills during locomotion of people who have suffered a moderate or severe head injury in the chronic phase in more ecological tasks. This will provide a better understanding of the difficulties encountered by these patients during locomotor interactions in everyday life.

ELIGIBILITY:
Inclusion Criteria for Traumatic Brain Injury group :

* 18 ≤ Age ≤ 55 years old
* Male/female
* Having suffered a first non-penetrating head injury
* Moderate to severe severity with initial Glasgow Coma Scale score 5<GCS<13
* In the subacute or chronic phase (≥ 3 months at the date of the experiment, relative to the date of the injury)
* Able to walk (10WMT speed ≥ 0.8 m/s, able to walk at least 20 m without technical or human assistance, PM ≥ 300 m)
* Able to maintain dynamic balance while standing (TUG<16s)
* Able to answer simple questionnaires, according to the investigator's judgment
* Having given their free, informed, expressed (written) consent
* Registered with a social security system
* Individuals under legal protection measures such as guardianship may be eligible

Inclusion Criteria for healthy control group :

* 18 ≤ Age ≤ 55 years old
* Male/female
* Able to walk (≥ 0.8 m/s, able to walk at least 20 m without technical or human assistance, PM ≥ 300 m)
* Able to answer simple questionnaires, according to the investigator's judgment
* Having given free, informed, expressed (written) consent
* Registered with a social security system

Exclusion Criteria specific to patients in the traumatic brain injury group :

- Person under legal protection (excluding guardianship) or unable to express consent

Exclusion Criteria for both groups :

* Severe patho-psychiatric care underway, which may impact the conduct of the protocol, at the investigator's discretion
* Presence of neurological signs suggestive of a neurodegenerative disease responsible for gait disturbance (Parkinson's syndrome, Alzheimer's disease, etc.)
* Individuals with musculoskeletal disorders that impact their locomotor abilities
* Presence of uncontrolled epilepsy at the time of inclusion
* Presence of visual impairments that make experimentation impossible, at the discretion of the investigator
* Pregnant, parturient, or breastfeeding women
* Participants in another ongoing research protocol involving human subjects

Exclusion Criteria for healthy control group :

* Presence of fatigue, trauma, or a condition affecting mobility, posture, balance, or walking
* Persons deprived of their liberty by a judicial or administrative decision
* Persons deprived of their liberty by judicial or administrative decision
* Persons under legal protection (guardianship, curatorship, judicial protection) or unable to express their consent
* Persons undergoing severe psychiatric treatment or admitted to a health or social care facility for purposes other than research.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Perceptive dimension : Elements of the environment viewed : Distribution (in %) | From enrollment to the end of the participation at maximum 30 days
Perceptive dimension : Elements of the environment viewed : Distance (in meters) | From enrollment to the end of the participation at maximum 30 days
Perceptive dimension : Elements of the environment viewed : duration of fixations (in milliseconds) | From enrollment to the end of the participation at maximum 30 days
Cognitive dimension : characteristics of the path taken : length of the path taken (in meters) | From enrollment to the end of the participation at maximum 30 days
Cognitive dimension : characteristics of the path taken : interpersonal distances with virtual humans (in m) | From enrollment to the end of the participation at maximum 30 days
Action-related dimension : walking speed (measured in m/s) | From enrollment to the end of the participation at maximum 30 days

SECONDARY OUTCOMES:
" Montréal Cognitive Assesment " (MoCA) | On day 1
" 10-Meter Walking Test " (10MWT) | At day 1
Balance test : ABC-scale | At day 1
Balance test : "Berg Balance Scale" (BBS) | At day 1
Balance test : "Time Up and Go" (TUG) | At day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Fondation Saint Helier, Rennes, France

IPD SHARING:
Plan to Share IPD: Undecided